CLINICAL TRIAL: NCT04434742
Title: The Effects of a Health-social Partnership Program for Discharged Non-frail Older Adults: a Pilot Study
Brief Title: The Effects of a Health-social Partnership Program for Discharged Non-frail Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Arkers, Wong, Clinical associate, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSP002
Record Dates: First submitted 2020-06-11; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Transition; Partner Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The subjects in this group receive complex interventions, including structured assessment, health education, goal empowerment, and care coordination supported by a health-social team.
  Interventions: Other: Complex interventions
- Control group (Other): The control group received usual discharge care and community resources that were made available to them as appropriate. A monthly social call was made to each client in the control group in order to exclude social effects. The contents of the social call, such as asking about entertainment and clients' hobbies, were set in the protocol.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Complex interventions — An advanced practice nurse (APN) from a hospital discharge team visited them to familiarize him/herself with their condition and prepare a discharge plan. A face-to-face or telephone call handover between the APN and the project nurse case manager (NCM) was performed before the client was discharged. The past and current medical conditions, medical and nursing management, and follow-up appointments were discussed. After discharge home, the NCM, functioning as the leader of health-social care team, conducted the initial assessment in the first home visit to identify the client's health and social problems within one week of discharge. Community workers, supervised by both the nurse case manager and social worker, provided telephone follow-up and subsequent home visits to monitor the client's progress and provide support when necessary.
  Arms: Intervention group
Other: Usual care — Social call was given to this group.
  Arms: Control group

SUMMARY:
Previous studies supporting discharged patients are hospital-based which admission criteria tend to include mainly those with complex needs and/or specific disease conditions. This study captured the service gap where these non-frail older patients might have no specific medical problem upon discharge but they might encounter residual health and social issues when returning home.

DETAILED DESCRIPTION:
Objective: To compare the effect of a community-based health-social partnership program with usual care for discharged community-dwelling non-frail older adults on their health-related quality of life, activities of daily living, depressive symptoms, and use of health services.

Design: A randomized controlled trial. Participants: Discharged community-dwelling non-frail older adults from an emergency medical ward in an intervention (n=37) and a control (n=38) group.

Interventions: Discharged older adults were randomized to receive usual care or complex interventions, including structured assessment, health education, goal empowerment, and care coordination supported by a health-social team.

Main measures: The outcomes were measured at pre-intervention (T1) and at three months post-intervention (T2) using the Medical Outcomes Study 12-item Short Form, the Modified Barthel Index and the Geriatric Depression Scale.

ELIGIBILITY:
Inclusion Criteria:

* resided in the service areas of the study hospital,
* were aged 60 or over,
* were cognitively competent with a score greater than 26 in the Montreal Cognitive Assessment Hong Kong version,
* were living at home before and after discharge from the hospital,
* had scores of <5 on the Clinical Frailty Scale (Note: a patient is considered to be non-frail if they have a score less than 5), and
* were fit for medical discharge

Exclusion Criteria:

* were not able to communicate,
* could not be reached by phone,
* were bed-bound,
* had active psychiatric problems,
* were already engaged in other structured health or social programs, and
* would not be staying in Hong Kong for the three months of the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Health-related quality of life: SF-12 at 3 months | At baseline pre-intervention and at three months when the interventions were completed.
  The goal for this program was to enable older adults to live with optimum quality of life in their own environment through receiving support from the collaboration of nurse case managers and social workers. Quality of life was measured by SF-12, which has been shown to be useful in Chinese elderly patients. The questionnaire has 12 items organized into eight categories (physical functioning, role limitation due to emotional and physical problems, mental health scale, general health, bodily pain, social functioning, and vitality), and has been validated in numerous studies.

SECONDARY OUTCOMES:
Change from baseline Activity of daily living at 3 months | At baseline pre-intervention and at three months when the interventions were completed.
  Use Modified Barthel index to measure the subjects' ability to do basic activity of daily livings such as grooming, eating, and walking. The score is from 0-100, with higher scores representing better activity of daily living.
Change from baseline Presence of depressive symptoms at 3 months | At baseline pre-intervention and at three months when the interventions were completed.
  The presence of depressive symptoms was measured by the Geriatric Depression Scale. The scores from each item are summed up. The maximum score is 15, with higher scores representing higher severity of depressive symptoms. Good validity and reliability have been reported in this scale, with criterion-related validity 0.95 and test-retest reliability 0.85 among the older Chinese population.
Change from Total number of unplanned outpatient department, general practitioner, and emergency department visits, hospital admissions and total number of health service attendances at 3 months | At baseline pre-intervention and at three months when the interventions were completed.
  This information was collected from the subjective reports of participants. They were asked about the number of attendances within the last three months prior to both T1 and T2 data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Arkers KC Wong, Dr, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Queen Elizabeth Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Wong AKC, Wong FKY, Ngai JSC, Hung SYK, Li WC. Effectiveness of a health-social partnership program for discharged non-frail older adults: a pilot study. BMC Geriatr. 2020 Sep 10;20(1):339. doi: 10.1186/s12877-020-01722-5. PMID 32912218